CLINICAL TRIAL: NCT07033234
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of HS-20118, and the Food Effect (FE) on the Pharmacokinetics in Adult Participants
Brief Title: Evaluate the Safety and Pharmacokinetics/Pharmacodynamics and Food Effect of HS-20118
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-20118-102
Record Dates: First submitted 2025-06-03; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20118 (Experimental): Single and multiple ascending doses of HS-20118 orally
  Interventions: Drug: HS-20118
- Placebo (Placebo Comparator): Single and multiple ascending doses of HS-20118-matched placebo orally
  Interventions: Drug: HS-20118

INTERVENTIONS:
Drug: HS-20118 — HS-20118

SUMMARY:
The study will be conducted in 2 parts (SAD and FE for Part 1 and MAD for Part2).

Part 1 is a single-center, randomized, double-blind, placebo-controlled, SAD study to evaluate the safety, tolerability, immunogenicity, and PK of HS-20118 and explore the food effect and fasting time on PK after a single oral dose in healthy participants.

Part 2 is a multi-center, randomized, double-blind, placebo-controlled, MAD study to evaluate the safety, tolerability, immunogenicity, PK, and PD of HS-20118 after multiple oral doses in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts (SAD and FE for Part 1 and MAD for Part2).

Part 1 is a single-center, randomized, double-blind, placebo-controlled, SAD study to evaluate the safety, tolerability, immunogenicity, and PK of HS-20118 and explore the food effect and fasting time on PK after a single oral dose after a single oral dose in healthy participants.

Part 1 will consist of 5 cohorts, i.e., X1 mg, X2 mg, X3 mg, X4 mg, and X5 mg dose cohorts (each cohort will include 3 participants to receive placebo). There will be no restriction on the male-to-female ratio. Each cohort will include 12 participants (HS-20118:placebo = 9:3), with a total of 60 participants. Participants will undergo PK blood sampling, ADA blood sampling, PD blood sampling and safety examinations during the study. It is planned to select a dose group in SAD to conduct a food effect study (to explore the possible effects of fasting time after taking the medicine and low-fat meals on HS-20118 PK).

Part 2 is a multi-center, randomized, double-blind, placebo-controlled, MAD study to evaluate the safety, tolerability, immunogenicity, PK, and PD of HS-20118 after multiple oral doses in patients with moderate to severe plaque psoriasis.

Part 2 will tentatively consist of 6 cohorts ( HS-20118 vs placebo = 9:3), i.e., (1) A1 mg, (2) A2 mg, (3) A3 mg, (4) A4 mg, (5) A5 mg, (6) A6 mg. Each cohort will include 12 participants (HS-20118:placebo = 9:3), with a total of 72 participants. There will be no restriction on the male-to-female ratio. Participants will undergo PK blood sampling, ADA blood sampling, PD blood sampling and safety examinations during the study.

ELIGIBILITY:
Inclusion Criteria:

For the SAD study:

1. Healthy adults aged 18-45 years (inclusive) at the time of signing the informed consent form;
2. Male participants weighing ≥ 50 kg and female participants weighing ≥ 45 kg, both ≤ 110 kg; body mass index (weight/square of height (kg/m2)) within the range of 18-28 kg/m2 (inclusive);
3. Normal results or abnormal results but without clinical significance in comprehensive examinations, including general physical examination, vital signs, laboratory tests, 12-lead ECG, abdominal color Doppler ultrasound, and chest X-ray from the frontal and lateral position ;

For the MAD study:

1. Male or female participants aged 18-65 years (inclusive) at the time of signing the informed consent form;
2. Male participants weighing ≥ 50 kg and female participants weighing ≥ 45 kg, both ≤ 110 kg;
3. Chronic plaque psoriasis for at least 6 months with or without psoriatic arthritis;

Exclusion Criteria:

For the SAD study:

1. Participants with immune-related diseases and medical history at screening;
2. Participants with a history of drug or other allergies who are considered by the investigator to be at high risk for participating in this study, or who may be allergic to the investigational medicinal product or any component of the investigational medicinal product as judged by the investigator;
3. History of drug abuse within the past 5 years or use of illicit drugs within 3 months before the study; or positive for urine drug screening;

For the MAD study:

1. Guttate psoriasis, pustular psoriasis, erythrodermic psoriasis, drug-induced psoriasis, or other diseases that affect the treatment results;
2. Current use of prohibited drugs or prior use of prohibited drugs within the specific time periods;
3. Known history of recurrent or chronic infections, or prior history of chronic or recurrent infections, including but not limited to: chronic renal infection, chronic chest infection (e.g., bronchiectasis), symptomatic urinary tract infection, and open, draining, or infected skin wounds; history of serious infections (e.g., sepsis, pneumonia, and pyelonephritis), or hospitalization or treatment with intravenous antibiotics for infections within 2 months before screening;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence, sever ity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation
Number of participants with abnormalities of physical examination | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Physical examination includes skin, mucous membranes, lymph nodes, head, neck, chest, abdomen, and spine/limbs, etc.
Number of participants with abnormalities of vital signs | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Vital sign measured include body temperature, blood pressure, pulse, and respiratory rate.
Number of participants with clinical laboratory abnormalities | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Clinical laboratory tests include blood biochemistry test, hematology test, urinalysis, coagulation function test, etc.
Number of participants with abnormalities of electrocardiogram (ECG) parameters | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  ECG parameters include heart rate, PR interval, RR interval, QRS duration, QTcF interval.

SECONDARY OUTCOMES:
Cmax | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Maximum plasma concentration
Tmax | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Time to reach Cmax
AUC | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Area under the plasma concentration-time curve
t½ | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Terminal half-life
CL/F | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Apparent clearance
Vd/F | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Apparent volume of distribution
Rac | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Accumulation ratio
Incidence of Anti-drug antibody (ADA) | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  Anti-drug antibody (ADA)
Proportions of psoriasis area and severity index (PASI) 75 | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The PASI assessment will assess erythema, thickening (plaque evaluation, induration), and scaling (desquamation) on the head, trunk, upper limbs, and lower limbs, respectively
Proportions of psoriasis area and severity index (PASI) 90 | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The PASI assessment will assess erythema, thickening (plaque evaluation, induration), and scaling (desquamation) on the head, trunk, upper limbs, and lower limbs, respectively
Proportions of psoriasis area and severity index (PASI) 100 | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The PASI assessment will assess erythema, thickening (plaque evaluation, induration), and scaling (desquamation) on the head, trunk, upper limbs, and lower limbs, respectively
Proportions of Investigator's Global Assessment (IGA) 0/1 | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The investigator scores each of infiltration/hypertrophy (I), erythema (E), and scaling (S) as a whole
Proportions of Investigator's Global Assessment (IGA) 0 | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The investigator scores each of infiltration/hypertrophy (I), erythema (E), and scaling (S) as a whole
Change from baseline in psoriasis area and severity index (PASI) total score | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The PASI assessment will assess erythema, thickening (plaque evaluation, induration), and scaling (desquamation) on the head, trunk, upper limbs, and lower limbs, respectively
Change from baseline in body surface area (BSA) | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The total BSA affected by plaque psoriasis is estimated based on the percent area affected, including head, trunk, upper extremities, and lower extremities
Change from baseline in dermatology life quality index (DLQI) | Day 1 up to Day 36 (SAD), Day 1 up to Day 71 (MAD)
  The DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne, and viral warts

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang, China